CLINICAL TRIAL: NCT06362057
Title: Biomechanical Effects of Digitally Constructed Subperiosteal Implants From Different Materials With Different Prosthetic Superstructures on Atrophied Maxilla: A Finite Element Analysis
Brief Title: Biomechanical Effects of Digitally Constructed Subperiosteal Implants
Status: Recruiting | Type: Observational
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, lecturer, Department of Prosthetic dental science, principle investigator, Menoufia University
Other Study IDs: 001-130125-017
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Bone Loss
Keywords: Polyetherketoneketone; Titanium; Polyethereetherketone
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Titanium framework group: Virtual design for Titanium subperiosteal framework group on atrophied maxilla.
  Interventions: Other: Subperiosteal implant framework
- PEEK framework group: Virtual design for PEEK subperiosteal framework group on atrophied maxilla.
  Interventions: Other: Subperiosteal implant framework
- PEKK framework group: Virtual design for PEKK subperiosteal framework group on atrophied maxilla.
  Interventions: Other: Subperiosteal implant framework

INTERVENTIONS:
Other: Subperiosteal implant framework — A 3D image of an edentulous maxilla bone will be derived from a computed tomography scan of an adult patient and saved as "stl" data. The solid geometry of the maxilla, including the cortical and spongious bone, was rebuilt from the "stl" data into the Digital Imaging and Communications in Medicine (DICOM) format with 3D-Doctor (Able Software Corp., MA, USA).
  With the Boolean method, force loading will be achieved between prosthetic parts, subperiosteal implant screws and bone tissues

SUMMARY:
Subperiosteal implants were first introduced in 1940 and then used worldwide for the treatment of edentulous maxilla or mandible with advanced bone atrophy.

DETAILED DESCRIPTION:
With the advancement of digital technology for the fabrication of materials and the emerging of new materials, subperiosteal implants can be fabricated from a wide variety of materials, and there is a lack of evidence regarding which material could be suitable.

ELIGIBILITY:
Inclusion Criteria:

* A 3D image of an edentulous maxilla bone derived from a computed tomography scan of an adult patient.
* Maxilla with Cawood and Howell class 4 or 5 classification

Exclusion Criteria:

* A 2D image of an edentulous maxilla bone
* A non atrophied maxilla

Ages: 30 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a three dimentional finite element analysis
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-07-27 (Estimated)

PRIMARY OUTCOMES:
bone loss under the implants | 10-15 years
  amount of bone loss which appears on a modeling process, The modeling process will be completed using a three-dimensional modeling software. A three-dimensional mesh consisting of 556,365 nodes and 2972,897 elements with VRMesh Studio (VirtualGrid Inc, Bellevue City, WA, USA) will used in the program.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A. El-Sawy, PhD, Study Chair — Menoufia University
Locations (1):
- Mohammed A. El-Sawy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
The IPD is upon request from the corresponding author

REFERENCES:
- [Derived] El-Sawy MA, El-Khatib B, Borg HS, Khater MT. Biomechanical effects of digitally constructed titanium, modified polyetheretherketone, and polyetherketoneketone subperiosteal implants on atrophied maxilla: a finite element analysis. BMC Oral Health. 2025 Jul 10;25(1):1142. doi: 10.1186/s12903-025-06426-z. PMID 40640731